CLINICAL TRIAL: NCT04430725
Title: Ablation of Lung Lesions Using Microwave Energy (ALLUME)
Brief Title: Microwave Ablation or Wedge Resection for the Treatment of Lung, Sarcoma and Colorectal Lesions, ALLUME Study
Status: Active, not recruiting | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 2018-0301; NCI-2020-03474 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2018-0301 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2020-06-10; First posted 2020-06-12 (Actual); Last update posted 2025-10-22 (Actual); Status verified 2025-10

CONDITIONS: Lung Non-Small Cell Carcinoma; Metastatic Colorectal Carcinoma; Metastatic Sarcoma; Stage I Lung Cancer AJCC v8; Stage IA1 Lung Cancer AJCC v8; Stage IA2 Lung Cancer AJCC v8; Stage IA3 Lung Cancer AJCC v8; Stage IB Lung Cancer AJCC v8; Stage II Lung Cancer AJCC v8; Stage IIA Lung Cancer AJCC v8; Stage IIB Lung Cancer AJCC v8; Stage III Lung Cancer AJCC v8; Stage IIIA Lung Cancer AJCC v8; Stage IIIB Lung Cancer AJCC v8; Stage IIIC Lung Cancer AJCC v8; Stage IV Colorectal Cancer AJCC v8; Stage IV Lung Cancer AJCC v8; Stage IVA Colorectal Cancer AJCC v8; Stage IVA Lung Cancer AJCC v8; Stage IVB Colorectal Cancer AJCC v8; Stage IVB Lung Cancer AJCC v8; Stage IVC Colorectal Cancer AJCC v8
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Colorectal Neoplasms; Sarcoma; Lung Neoplasms | interventions — Contrast Media; Microwaves

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Tissue
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Observational (microwave ablation, wedge excision, CT): Patients undergo standard care microwave ablation or wedge resection followed by contrast-enhanced CT imaging at 1, 6, 12, 18 and 24 months. Patients also complete questionnaires over 10-15 minutes at baseline up to 9 months.
  Interventions: Procedure: Computed Tomography with Contrast; Procedure: Microwave Ablation; Other: Questionnaire Administration; Procedure: Wedge Excision

INTERVENTIONS:
Procedure: Computed Tomography with Contrast — Undergo contrast-enhanced CT
  Other Names: Contrast Enhanced Computed Tomography; CONTRAST ENHANCED CT SCAN; Contrast-enhanced Computed Tomography; CT Scan With Contrast; CT with Contrast
Procedure: Microwave Ablation — Undergo microwave ablation
  Other Names: Ablation, Microwave
Other: Questionnaire Administration — Ancillary studies
Procedure: Wedge Excision — Undergo wedge resection
  Other Names: Wedge Resection

SUMMARY:
This study compares the outcomes and safety of two standard treatment options called microwave ablation and surgical wedge resection in patients with non-small cell lung cancer, sarcoma and colorectal cancer that has spread to other parts of the body (metastatic). Microwave ablation is designed to kill tumor cells by heating the tumor until the tumor cells die. A wedge resection is a procedure that involves the surgical removal of a small, wedge-shaped piece of lung tissue to remove a small tumor or to diagnose lung cancer. Comparing these two treatment options may help researchers learn which method works better for the treatment of non-small cell lung cancer, metastatic sarcoma, and metastatic colorectal cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. Estimate the 2-year local recurrence rate for microwave ablation within a basket.

SECONDARY OBJECTIVES:

I. Evaluate whether microwave ablation offers treatment benefit for safety when compared to wedge resection using a contemporaneous database consisting of a commensurate surgical patient population.

II. Evaluate whether microwave ablation offers treatment benefit for efficacy when compared to wedge resection using a contemporaneous database consisting of a commensurate surgical patient population.

III. Evaluate whether microwave ablation offers treatment benefit for changes in patient reported outcomes when compared to wedge resection using a contemporaneous database consisting of a commensurate surgical patient population.

OUTLINE:

Patients undergo standard care microwave ablation or wedge resection followed by contrast-enhanced computed tomography (CT) imaging at 1, 6, 12, 18 and 24 months. Patients also complete questionnaires over 10-15 minutes at baseline up to 9 months.

ELIGIBILITY:
Inclusion Criteria:

* Patient has a lung lesion(s) that is either biopsy-proven cancer or shows sequential growth on CT imaging with clinical suspicion for non-small cell lung cancer (NSCLC)-stage I; NSCLC-stage > 1; metastatic sarcoma; or metastatic colorectal (CRC) cancer
* 3 cm or less tumor size
* Other sites for cancer are either controlled or there are plans for control
* Expected margin at least 1 cm from critical structures, allowing for protective strategies such as induction of therapeutic pneumothorax. Critical structures include the trachea, main bronchi, esophagus, aorta, aortic arch branches, superior vena cava (SVC), main, right or left pulmonary artery, or heart.

Exclusion Criteria:

* Patient is considered high risk for ablation due to major comorbid medical conditions
* Patient is pregnant or breast feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with non-small cell lung cancer, metastatic sarcoma, or metastatic colorectal cancer.
Sampling Method: Non-Probability Sample
Enrollment: 74 (Actual)
Dates: Start 2019-08-07 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
Time to local recurrence per treated nodule | Up to 2 years post-ablation
  Will be measured from the first date of treatment and characterized according to the Response Evaluation Criteria in Solid Tumors (RECIST) criteria and/or biopsy. The local recurrence of each subtype will be adjusted according to the method proposed by Fine and Gray. Will evaluate each basket individually and allow patients to contribute multiple nodules. Therefore, the Bayesian piecewise constant frailty model will be used to account for interdependence in the failure duration of nodules arising from the same patient. Additional posterior summaries will be reported, such as median failure duration. Additionally, will report plots of the full time-to-failure distribution with pointwise 95% Bayesian credible intervals.

SECONDARY OUTCOMES:
Incidence of clinically significant adverse events | Up to 30 days
  The occurrence of significant adverse events will be recorded according to the Common Terminology Criteria for Adverse Events (CTCAE) published by the National Institutes of Health. Grade III or above adverse events within the following categories: cardiac disorders, general disorders and administration site conditions, infections and infestations, injury, poisoning and procedural complications, and respiratory, thoracic and mediastinal disorders. 30-day mortality will also be recorded. Patient adverse events will be tabulated by symptom grade and categories.
Time to local recurrence per patient | Up to 2 years post-ablation
  Contrast-enhanced CT imaging will be used to monitor for local recurrence. Local recurrence will be defined either by a positive biopsy or by radiographic RECIST criteria. Frequentist interference will use the Kaplan-Meier method.
Regional and distance recurrence | Up to 2 years post-ablation
  Regional and distant recurrence will be defined either by a positive biopsy or by radiographic RECIST criteria. Frequentist interference will use the Kaplan-Meier method.
Overall survival per patient | Up to 2 years post-ablation
  Frequentist interference will use the Kaplan-Meier method.
Changes in patient reported outcomes per patient | Up to 9 months after enrollment
  Will be reported as time to symptom recovering using MD Anderson Symptom Inventory-Lung Cancer (MDASI-LC) questionnaires. Frequentist interference will use the Kaplan-Meier method.

CONTACTS AND LOCATIONS:
Overall Officials: Wayne L Hofstetter, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org